CLINICAL TRIAL: NCT03244293
Title: Sensitivity and Specificity of Bispectral Index (BIS) for Classification of Procalcitonin (PCT) Sepsis Grades in Critically Ill Patients With Sepsis, Severe Sepsis and Septic Shock and Multiple Organ Failure (MOF)
Brief Title: Bispectral Index (BIS) for Classification of Procalcitonin (PCT) Sepsis Grades in Critically Ill Patients With Sepsis
Acronym: BIS6
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Ashraf A. Dahaba, Principle Investigator, Suez Canal University
Other Study IDs: MUGraz6
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Sepsis, Severe
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
To evaluate the discriminative power of BIS monitoring to classify the degree of mental state associated with the PCT graded sepsis cascade, and to assess its utility for monitoring the improvement or deterioration of sepsis.

DETAILED DESCRIPTION:
To evaluate the discriminative power of BIS monitoring to classify the degree of mental state associated with the PCT graded sepsis cascade, and to assess its utility for monitoring the improvement or deterioration of sepsis. The primary endpoint of our study was to use an artefact-free 10-min mean BIS value to classify the degree of sepsis. As secondary endpoints, we correlated the mean BIS value to various mental state and sepsis parameters; PCT, C-reactive protein (CRP), Glasgow coma scale, and sequential organ failure assessment (SOFA) score. In a longitudinal study, patients' PCT sepsis grades were reassessed at a later time point and a second artefact-free 10-min mean BIS value was recorded to evaluate BIS evolution within the same patient.

ELIGIBILITY:
Inclusion Criteria: patients with sepsis

* patients with sepsis

Exclusion Criteria:

* Patients who received drugs that would interfere with BIS monitoring

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critical Care patients with all grades of Sepsis monitored with bispectral index
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Bispectral Index (BIS)-Electroencephalography (EEG) derived parameter correlated to the severity of Sepsis as indicated by Procalcitonin (PCT) biomarker. | Time point 1= On CCU admission, Time point 2= day 3 of CCU admission, Time point 3= on release from CCU.
  Bispectral Index (BIS)-Electroencephalography (EEG) derived parameter (scale from 0=brain dead to 100= normal EEG) will be monitored and correlated to the severity of Sepsis as indicated by daily measured Procalcitonin (PCT) biomarker (<0.5 micg/L =no sepsis up to 100 micg/L =Septic shock)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Dahaba, MD, MSc, Principal Investigator — Suez Canal University
Locations (1):
- Dalian Medical University, Dalian, Dalian, China

IPD SHARING:
Plan to Share IPD: No